CLINICAL TRIAL: NCT04411290
Title: Correlation of Malignancy Predictors, Bethesda (I-VI) and TI-RADS Scores (I-V) With Final Histopathology in Patients Undergoing Total Thyroidectomy 34 Years After Chernobyl Disaster: Multi-centric Trial
Brief Title: Malignancy Predictors, Bethesda and TI-RADS Scores Correlated With Final Histopathology in Thyroid Diseases
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ethem Unal, M.D., PhD, Associate Prof of Surgery & Surgic, Assoc. Professor of General Surgery and Surgical Oncology, Umraniye Education and Research Hospital
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/172
Record Dates: First submitted 2020-05-15; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Thyroid Carcinoma; Thyroid Papillary Carcinoma; Multinodular Goiter, Adolescent; Solitary Thyroid Nodule; Thyroid Diseases; Multifocal Dysplasia; Aspiration; Thyroid Nodule; Thyroid Cancer, Papillary; Thyroid Neoplasms; Thyroid Goiter
Keywords: Total Thyroidectomy; Black Sea; Eastern Europe; Radiation; Endemic; Fine needle aspiration (FNA); Multifocality; Bethesda; Cytology; Thyroid Imaging Reporting and Data System (TI-RADS); International; Multi-centric; Multicentric study
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary; Euthyroid Goiter; Thyroid Diseases; Thyroid Nodule; Goiter; Burkitt Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Thyroidectomy (TT)-indicated patients: Patients with presumably benign thyroid disease (multinodular goitre, solitary thyroid nodule, toxic goitre, etc.) Patients with thyroid carcinoma (biopsy-proved) Total thyroidectomy preference by the primary surgeon
  Interventions: Procedure: Total thyroidectomy (TT)

INTERVENTIONS:
Procedure: Total thyroidectomy (TT) — Final total thyroidectomy histopathology report should be available for correlations with preoperatively determined malignancy predictive factors, Bethesda (cytology) and TI-RADS (ultrasound findings)

SUMMARY:
In the last decades, thyroid cancer incidence has continuously increased all over the world, almost exclusively due to a sharp rise in the incidence of the papillary histologic subtype, which has the highest incidence of multifocality. Furthermore, Black Sea and Eastern European regions are both endemic and known to have been under the influence of Chernobyl nuclear explosion. Although overscreening might have a role in certain parts of the world, the predictors of malignancy such as family history, genetical disorders, previous radiation exposure, low iodine intake, diabetes and obesity, should also be taken into consideration in determining the extent of surgery.

DETAILED DESCRIPTION:
High-frequency ultrasound (US) is increasingly used to help distinguish malignancy in patients with solitary or multiple nodules, and US-guided fine needle aspiration (FNA) has become the gold standard test for detecting thyroid cancer. Moreover, a further US-based risk stratification of thyroid nodules with Thyroid Imaging Reporting and Data System (TI-RADS) has been currently proposed for better and easier decision making. However, the presence of multiple nodules in the thyroid gland may decrease the diagnostic value of these preoperative diagnostic tools. The prevalence of incidental carcinoma identified on the final histological examination of the patients who underwent surgery for presumably benign thyroid diseases was previously reported to be roughly around 5 to 10%. Most of the previous studies also showed a lower risk of carcinoma in multinodular goitre (MNG) compared to solitary thyroid nodule (STN). However, some recent surgical series have reported that the risk of thyroid carcinoma in benign thyroid diseases is significantly higher than previously reported.

The purpose of the present study is to detect the accuracy of preoperative cytology and US-findings (TI-RADS) and the prevalence of thyroid carcinoma in patients operated for thyroid diseases and to discuss all malignancy risk factors in detail along with final histopathological report. Cytology-histology discrepant cases will also be further evaluated for sampling and interpretation errors, and possible solutions to increase the accuracy of preop testing are going to be proposed. The accuracy of the preference of total thyroidectomy procedure will be evaluated considering the prevalence of incidental carcinomas diagnosed postoperatively, and whether there are variations in the risk of malignancy with respect to final pathology of patients will also be discussed in detail.

ELIGIBILITY:
Inclusion Criteria:

* >17 years all patients with benign/malign thyroid disease, total thyroidectomy is indicated/preferred by both primary surgeon and patient (signed informed consent is a must)
* All patients should have a malignancy predictive factors forms filled in
* All patients should have fine needle aspiration cytology (Bethesda category) available
* All patients should have an ultrasound evaluated according to TI-RADS
* All patients should have a final histopathology report

Exclusion Criteria:

* Patients who are prepared for thyroid surgery other than total thyroidectomy procedure
* Age<17 years

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with benign or malign thyroid disease, eligable for total thyroidectomy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative Evaluation of Malignancy Risk Factors-How many risk factors are present? | 12 months
  Malignancy risk factors: 1. Demographics (Age and gender-Male/Female), 2. Smoking history (Yes/No, duration and number/day), 3. Iodine-deficient diet (Yes/No), 4. Born at an endemic area (Yes/No), 5. Presence in an endemic area (Yes/No), 6. Radiation exposure (Yes/No), 7. Radiation treatment during childhood (Yes/No), 8. Head and neck carcinoma (Yes/No), 9. Other carcinoma history (Yes/No, if yes specify.........) 10. Family history of thyroid disease (Yes/No), 11. Family history of other carcinomas (Yes/No), 12. Personal history of thyroid carcinoma/surgery (Yes/No, if yes, pathology……..), 13. Personal history of other carcinomas (e.g. colonic polyps? breast disease?......) 14. Genetic disorders (Yes/No), 15. Obesity (Body mass index - ? kg/m2), 16. Diabetes mellitus (Yes/No) should be evaluated for each patient before surgery- The number of risk factors will be compared with malignancy rate found at final histopathology report.
Preoperative Bethesda category, Fine needle aspiration (FNA) cytology report | 12 months
  Bethesda score-FNA cytology report- as I, II, III, IV, V or VI. Cytology report will be compared with final histology report for each patient for malşgnancy rate and multifocality I. Nondiagnostic or unsatisfactory, II. Benign, III. Atypia of undetermined significance (AUS) or follicular lesion of undetermined significance (FLUS), IV. Follicular neoplasm or suspicious for a follicular neoplasm-Preoperative cytology category will be compared with postoperative final histopathology report for malignancy rate, multifocality and cases with cytology-histopathology discrepancy will be evaluated further for biopsy techniques and cytology mis-interpretations.
  V. Suspicious for malignancy, VI. Malignant.
Preoperative ultrasound evaluation with Thyroid Imaging Reporting and Data System (TI-RADS) | 12 months
  TI-RADS score-Ultrasound evaluation of thyroid nodues- as I, II, III, IV or V. TI-RADS scores will be compared with final histopathology report to see malignancy rates and accuracy of TI-RADS.
  TI-RADS 1: Normal thyroid gland. No focal lesion. TI-RADS 2: Benign nodules. Noticeably benign pattern (0% risk of malignancy) TI-RADS 3: Probably benign nodules (<5% risk of malignancy)
  TI-RADS 4:
  * 4a - Undetermined nodules (5-10% risk of malignancy) Score of 1.
  * 4b - Suspicious nodules (10-50% risk of malignancy) Score of 2.
  * 4c - Highly suspicious nodules (50-85% risk of malignancy) Score of 3-4 TI-RADS 5: Probably malignant nodules (>85% risk of malignancy) Score of 5 or higher TI-RADS 6: Biopsy-proven malignancy
Total thyroidectomy for both benign and malign thyroid diseases | 12 months
  Final histopathology report-After surgery (all patients should have a final histopathology report after total thyroidectomy operation). Final histology report will be correlated to Malignancy risk factors (number), Bethesda category (accuracy, false negativity/positivity) and TI-RADS (accuracy, false negativity/positivity)

CONTACTS AND LOCATIONS:
Overall Officials: Ethem UNAL, MD, PhD, Study Chair — Assoc. Professor of General Surgery and Surgical Oncology; Sema YUKSEKDAG, MD, Principal Investigator — Instructor in General Surgery
Locations (1):
- Umraniye Education and Research Hospital, Health Sciences Universit, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All Excel documents will be available (Patient initials and medical record numbers shaded XX). Demographics, BMI, malignancy risk factors, Bethesda and TI-RADS scores and final histopathology reports
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: June 01, 2020
Access Criteria: Contact for all available forms by email Open to all centers (especially for Black Sea and Estern European centers, but not limited to)

REFERENCES:
- [Result] Delfim RLC, Veiga LCGD, Vidal APA, Lopes FPPL, Vaisman M, Teixeira PFDS. Likelihood of malignancy in thyroid nodules according to a proposed Thyroid Imaging Reporting and Data System (TI-RADS) classification merging suspicious and benign ultrasound features. Arch Endocrinol Metab. 2017 May-Jun;61(3):211-221. doi: 10.1590/2359-3997000000262. Epub 2017 Mar 27. PMID 28699990
- [Result] Tufano RP, Noureldine SI, Angelos P. Incidental thyroid nodules and thyroid cancer: considerations before determining management. JAMA Otolaryngol Head Neck Surg. 2015 Jun;141(6):566-72. doi: 10.1001/jamaoto.2015.0647. PMID 25928353
- [Result] Tan H, Li Z, Li N, Qian J, Fan F, Zhong H, Feng J, Xu H, Li Z. Thyroid imaging reporting and data system combined with Bethesda classification in qualitative thyroid nodule diagnosis. Medicine (Baltimore). 2019 Dec;98(50):e18320. doi: 10.1097/MD.0000000000018320. PMID 31852120
- Available data/document: Principal investigator data — https://scholar.google.com.tr/citations?user=6bFlCZwAAAAJ&hl=tr